CLINICAL TRIAL: NCT02387593
Title: Usefulness of Endocuff in the Adenoma Detection Rate. A Randomized Clinical Trial
Brief Title: Usefulness of Endocuff in the Adenoma Detection Rate. Comparative Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Dr. Rafael Barreto Zúñiga, Attached to the Department of Endoscopy Medical Institute, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: END-1302-14/15-1
Record Dates: First submitted 2015-03-09; First posted 2015-03-13 (Estimated); Last update posted 2015-03-13 (Estimated); Status verified 2014-09

CONDITIONS: Colorectal Canceer
Keywords: Adenoma; Colonoscopy; Screening
MeSH Terms: conditions — Adenoma

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- colonoscopy with endocuff (Experimental): To the usual colonoscopy will place a endocuff at the tip of the colonoscope
  Interventions: Device: ENDOCUFF
- standard colonoscopy without endocuff (No Intervention): Routine colonoscopy without endocuff

INTERVENTIONS:
Device: ENDOCUFF — One endocuff device is placed at the tip of colonoscope prior to colonoscopy baseline
  Arms: colonoscopy with endocuff

SUMMARY:
Colorectal cancer (CRC) is one of the leading causes of cancer death worldwide. The cumulative risk of developing CRC is about 6% lifelong.

The benefit of screening colonoscopy depends on the detection and removal of all adenomas, however, some of these may be difficult to detect.

The "endocuff" (EC) is a polymer sleeve which joins the tip of the colonoscope to improve the image viewing of the mucosa during colonoscopy procedure.

There is insufficient evidence of the usefulness of endocuf

DETAILED DESCRIPTION:
All patients requiring colonoscopy for screening and who agree to participate in the study will be included and randomized them to make an standard colonoscopy or colonoscopy with endocuff, for randomization system will be used in balanced blocks of 4, created on the page randomization.com.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult patients,
* Aged 18,
* Who would come to colonoscopy for colon cancer screening without prior colonoscopy studies

Exclusion Criteria:

* Boston colonic preparation <5 points
* Suspected Lynch syndrome or familial adenomatous polyposis (FAP)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Adenoma detection rate | 30 minutes
  Percentage of adenomas detected during colonoscopy
Measurement of the polyp detection rate | 30 minutes
  Percentage of polyps detected during colonoscopy

SECONDARY OUTCOMES:
Cecal intubation rate | 30 minutes
  Percentage of cecal intubation
ileal intubation rate | 10 minutes
  Percentage of ileal intubation
Difficulty performing polypectomy | 10 minutes
  When the endoscopist requiring special maneuvers to perform polypectomy
Complications during colonoscopy | One week
  When patients require special handling during or immediately subsequent colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Rafael, MD, Principal Investigator — Department of Endoscopy
Locations (1):
- Rafael Barreto, México, Tlalpan, Mexico